CLINICAL TRIAL: NCT03494621
Title: A CBPR Initiative for Reducing Infant Mortality In American Indian Communities
Brief Title: Infant Care Practices Study
Acronym: ICP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017088; R01HD080544-01 (NIH)
Record Dates: First submitted 2018-03-19; First posted 2018-04-11 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Sudden Infant Death
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants randomly assigned to the control group will have three prenatal contacts at the same gestational ages as the intervention participants. These contacts will include collection of covariate data, review of locally available educational materials on pregnancy/infant care led by trained study staff, and assessment of the overall session quality and acceptability. The educational materials provided during these sessions are drawn from materials currently available at local health care facilities
- Protecting Babies While They Sleep (Experimental): The intervention curriculum derives from information gathered at previously conducted focus groups and interviews, which aimed to ascertain the role of caregiver knowledge, beliefs, and access to resources in implementation of infant safe sleep practices. The protocol for the focus groups and interviews has been reviewed by the Tribal Institutional Review Board. The focus groups were conducted in Rapid City and a western Tribal reservation with pregnant adult women and pregnant, parenting, or other interested adolescent women; fathers (adult men); and elder women. Two focus groups were held for each category of individuals. Additional qualitative data was collected via key informant interviews with individuals vested and experienced in maternal and child health.
  Interventions: Behavioral: Protecting Babies While they Sleep Curriculum

INTERVENTIONS:
Behavioral: Protecting Babies While they Sleep Curriculum — The intervention curriculum derives from information gathered at previously conducted focus groups and interviews, which aimed to ascertain the role of caregiver knowledge, beliefs, and access to resources in implementation of infant safe sleep practices. .
  Arms: Protecting Babies While They Sleep

SUMMARY:
This proposed project will engage American Indian communities through existing partnerships, utilizing a Community Based Participatory Research (CBPR) methodology to design a group intervention program to increase the safety of infant sleep environments. Compelling evidence from research in other racial populations suggests that family and cultural norms, attitudes and personal beliefs about infant sleep, safety and comfort are strongly associated with the choice of infant sleep environment. It may be possible that the current safe sleep messages are in conflict with inherent cultural beliefs within these communities. This conflict with the scientific recommendations regarding safe sleep may influence behavior, even in the presence of adequate knowledge about safe sleep practices. Preliminary discussions with many tribal leaders and elders suggest that this chasm between culture and scientific recommendations can be bridged with an intervention incorporating culture, education and resources. However, there is limited research on factors influencing infant safe sleep practices of American Indian mothers. This study will test the effectiveness of incorporating cultural beliefs and practices into an intervention package based on the American Academy of Pediatrics safe sleep guidelines that incorporates both education and provision of resources. Therefore, the research question is: "Does a culturally specific safe sleep intervention, developed using CBPR, reduce the risk of unsafe infant sleep practices in Northern Plains American Indian communities?"

DETAILED DESCRIPTION:
The proposed study is a two-group randomized trial with a total sample size of 150. Pregnant women from Western South Dakota who meet eligibility criteria will be randomly assigned to an intervention or a control group and will be followed through their pregnancy and postnatal period until their infant reaches one year of age. They will remain in their randomized group throughout the course of the study.

Intervention group: Participants randomly assigned to the intervention group will have three prenatal contacts at study site offices. These contacts will include collection of covariate data, engagement with the Protecting Babies While They Sleep curriculum and activities (described below) led by trained study staff, and assessment of the overall session quality and acceptability. Participants will be allowed to invite up to two family members or other support persons to attend the third prenatal contact. The research coordinator will review the consent form and request consent for each guest of the participant. Guests will be asked to provide a subset of the covariate data provided by the primary participant, engage with the curriculum and associated activities, and assess the overall session quality and acceptability.

The intervention curriculum derives from information gathered at previously conducted focus groups and interviews, which aimed to ascertain the role of caregiver knowledge, beliefs, and access to resources in implementation of infant safe sleep practices. The study investigators worked with a Community Advisory Board (CAB) to design the focus group and interview questions, interpret the resulting qualitative data, and guide development of the intervention curriculum. The curriculum combines culturally-based prenatal and infant care education with current safe sleep recommendations from the American Academy of Pediatrics (AAP). The main components include: brief videos featuring medical professionals and American Indian elders, discussion guided by Motivational Interviewing principles, and culturally-based activities designed to reinforce the curriculum objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identified as American Indian
2. Able to provide informed consent or assent
3. Mother's age 14 years or older
4. If emancipated minor, not living in group home or care facility
5. Gestational age 20 weeks or less
6. No planned relocation outside the catchment area
7. Fluency in English

Exclusion Criteria:

1. Not self-identified as American Indian
2. Unable to provide informed consent or assent
3. Mother's age less than 14 years
4. Emancipated minor living in group home or care facility
5. Gestational age more than 20 weeks
6. Planned relocation outside of the catchment area
7. Not fluent in English

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Yes
Enrollment: 115 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Implementation of safe sleeping practices | Three months
  Primary outcome will be measured by participant report about infant sleep location and sleep position. Infant location is considered safe if participant reports a 'no' response to if the participant shared a sleep location with baby. INfant sleep position is considered safe if the participant provides a 'yes' response to whether the baby was put on its back to sleep for every sleep. The two responses will be aggregated together to derive that the participant is practicing safe sleep habits.If either question indicates unsafe sleeping habits, the participant will be counted as not practicing safe sleeping habits.

SECONDARY OUTCOMES:
Change in Safe Sleep knowledge | prenatal, 3 months postnatal, 6 months postnatal, 1 year
  The impact of the intervention on the participant's knowledge of safe sleep will be assessed through participant self report.
Change in beliefs regarding infant safe sleep | prenatal, 3 months postnatal, 6 months postnatal, 1 year
  The impact of the intervention on the participants' belief regarding infant safe sleep will be measured through self report
Change in safe sleep practice | prenatal, 3 months postnatal, 6 months postnatal, 1 year
  The impact of the intervention on the participants' practice of safe sleep will be measured through self report

CONTACTS AND LOCATIONS:
Overall Officials: Amy Elliott, PhD, Principal Investigator — Avera Research Institute
Locations (1):
- Avera Research Institute, Rapid City, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators understand that sharing of research data with the broad research community promotes collaboration and further development of the scientific field. The investigators intend to share de-identified data with NIH in accordance with tribal policies and regulations. The investigators anticipate that a detailed plan will be in place to allow for sharing of data after analysis and publication of the primary hypothesis.

DOCUMENTS (1):
  • Informed Consent Form (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT03494621/ICF_001.pdf